CLINICAL TRIAL: NCT05013541
Title: Effect of Bladder Filling on Rectal Contractions During Cystometry
Status: Completed | Type: Observational
Sponsor: Gérard Amarenco (Other)
Responsible Party: Sponsor-Investigator, Gérard Amarenco, Head of Neuro-Urology department, Tenon Hospital, Pierre and Marie Curie University
Organization: Pierre and Marie Curie University (Other)
Other Study IDs: GREENGRC01
Record Dates: First submitted 2021-08-16; First posted 2021-08-19 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Bladder Dysfunction
Keywords: urodynamics; rectum / physiopathology; muscle contraction / physiology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients included: Patients with lower urinary tract disorders assessed with multichannel cystometry and presence of rectal contractions.
  Measure of amplitude and frequency of rectal contractions function of the bladder sensation and volume of bladder filling.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Observational study, standard record of need to void during cystometry

SUMMARY:
Increasing knowledge on rectal motility and bladder-rectum cross-talk has been published in recent years. However, whether bladder filling factors during multichannel urodynamic studies affect rectal contraction (RC) parameters has not been studied.

The primary aim of this study is to assess the impact of bladder filling and desire to void on rectal contraction amplitude or frequency.

Secondary objectives are to determine any significant change in rectal parameters depending on clinical and urodynamic factors or treatment.

All patients referred for urodynamic assessment and with studies positive for rectal contractions as defined by the international continence society (ICS) will be included. Abdominal pressure will be measured using a T-doc air charged abdominal catheter inserted 10 cm from the anal margin. Standardized urodynamic evaluation will be conducted following ICS guidelines.

Mean amplitude, maximal amplitude (cmH20) and mean frequency of rectal contractions on all urodynamic studies will be visually measured on the recording software and compared depending on bladder sensation (First Desire to void (FDV), Strong Desire to Void (SDV) and filling volume (200ml, 400ml).

Demographic data (age, sex, BMI), underlying neurological disease, clinical symptoms, and scores (Neurogenic Bladder Symptom Score, Bristol Score, Cleveland Score), urodynamic parameters and treatments will be collected. Time since last defecation and meal will also be collected.

This prospective observational study will be conducted in a Neuro-Urology department of a French university hospital. All the patients included are referred for multichannel urodynamic assessment.

DETAILED DESCRIPTION:
Studies have suggested multiple types of colonic motor patterns including rectal motor activity. This rectal activity has been described in conventional multichannel urodynamic studies and has been determined not be an artefact. Some studies have related this rectal activity to bladder dysfunction, an underlying neurological affection or old ageing. However, the significance of this rectal activity observed during urodynamic studies remains unclear. It has been suggested that rectal activity may be a marker for underlying conditions.

On the other hand, rectal phasic contractions using conventional manometry have been described for decades and consecutively coined rectal motor activity, periodic rectal motor activity and rectal motor complex. Recent data using High Resolution Manometry reports retrograde propagating cyclic motor patterns occurring with a frequency of 2 to 6 events per minute. In this study 59% of retrograde CMPs initiated in the sigmoid colon and rectum in the postprandial period suggesting a mechanism to limit rectal filling. This supports Rao and al.'s theory of a rectosigmoid brake. Modifications of CMP have also been shown in pathology such as slow transit constipation and fecal incontinence although results are conflicting.

Furthermore, rectum and bladder share a common embryological origin and innervation which has led in recent years to the development of the concept of a cross talk between rectum and bladder. Animal and human studies have assessed the effect of rectal distension on bladder sensation and motility. However, whether bladder filling factors affect rectal contraction parameters has not been specifically studied.

The primary aim of this study is to assess if bladder sensation and filling volume have any significant effect on rectal contraction parameters such as amplitude or frequency. Secondary objectives are to determine any significant change in rectal parameters depending on clinical and urodynamic factors or treatment.

This prospective observational study will be conducted in a Neuro-Urology department of a French university hospital. All the patients included are referred for multichannel urodynamic assessment to explore urinary disorders.

All patients referred for urodynamic assessment will be screened. All patients with a recording of rectal contractions as defined by the international continence society (ICS) during the urodynamic study will be included. Rectal contraction identified by a first investigator will have to be confirmed by a second investigator to be included for further analysis. The ICS defines rectal contractions as: temporary phasic increases in abdominal pressure without synchronous change in vesical pressure resulting in negative deflections of detrusor pressure. Based on previously published studies, rectal contractions resulting in a more than 5 cmH20 change of abdominal pressure will be included for analysis. Abdominal pressure will be measured using a T-doc air charged abdominal catheter inserted 10 cm from the anal margin. Patients will be informed on the procedure prior to the exam. Filling of the bladder will be carried out in a semi-seated position. Patients will be asked to report need to void; FSF, First Desire to Void (FDV) and SDV.

The following data will be collected: age, sex, body mass index, etiology of urinary disorders, type of urinary or bowel symptoms, use of treatment for urinary or bowel dysfunction, time of last meal, detrusor overactivity on urodynamics.

Amplitude and frequency of rectal contractions will be measured individually on the software used for the urodynamic study. The amplitude of each contraction will be measured as the difference between the peak of the contraction wave and the baseline preceding each contraction. Mean and maximum amplitude will be compared between time samples depending on bladder sensation and filling volume. The frequency will be calculate as (number of contraction on the studied period)/(time of the studied period). Absence of contraction on a sample will be counted as a frequency of 0. The occurrence of at least 2 contractions over a time sample will be necessary in order for an average frequency to be calculated. Frequency of contractions will be compared between beginning of cystometry to first desire to void (FDV) and FDV to end of bladder filling.

Secondary analysis to assess the impact of clinical and urodynamic data on rectal contraction parameters will be performed.

All data will be collected and analyzed without any identifying information.

ELIGIBILITY:
Inclusion Criteria:

* age over 18
* lower urinary tract dysfunction requiring cystometry assessement
* rectal contraction during cystometry

Exclusion Criteria:

* Colo-rectal inflammatory or oncological disease
* History of colo-rectal surgery
* Irritable bowel syndrome
* Probe expulsion (during urodynamic study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: observational cohort of included patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Variation of the amplitude of rectal contraction function of bladder sensation 1 | One day
  Difference of mean amplitude of rectal contraction between beginning of cystometry to first desire to void (FDV) and FDV to end of bladder filling (maximal capacity)

SECONDARY OUTCOMES:
Variation of the amplitude of rectal contraction function of bladder sensation 2 | one day
  Difference of mean amplitude of rectal contraction between beginning of cystometry to first desire to void (FDV) and FDV to Strong Desire to Void (SDV)
Variation of the amplitude of rectal contraction function of bladder sensation 3 | One day
  Difference of maximal amplitude of rectal contraction between beginning of cystometry to first desire to void (FDV) and FDV to end of bladder filling (maximal capacity)
Variation of the amplitude of rectal contraction function of bladder sensation 4 | One day
  Difference of maximal amplitude of rectal contraction between beginning of cystometry to first desire to void (FDV) and FDV to Strong Desire to Void (SDV)
Frequency of rectal contraction function of bladder sensation | One day
  Difference of mean frequency of rectal contraction between beginning of cystometry to first desire to void (FDV) and FDV to end of bladder filling
Variation of the amplitude of rectal contraction function of bladder filling | One day
  Difference of mean amplitude of rectal contraction between beginning of cystometry to 200mL of bladder filling and 200 to 400mL of bladder filling (maximal capacity)
Rectal contraction parameters function of patients' characteristics | One day
  Difference of rectal contraction parameters (Mean amplitude, maximal amplitude and frequency) depending on demographic data (age, sex, BMI), underlying neurological disease, clinical symptoms, urodynamic status and treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Gérard Amarenco, PUPH, Principal Investigator — Sorbonne Université, GRC 001, GREEN, AP-HP, Hôpital Tenon, Paris, France
Locations (1):
- department of Neuro-Urology, Hôpital Teno, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided